CLINICAL TRIAL: NCT01575613
Title: Reducing the Burden of Malaria by Targeting Hotspots of Transmission and Improving Malaria Control Measures in the Highlands of Western Kenya: Simultaneous Rollout of Four Malaria Control Interventions and Evaluation by Cross-sectional Surveys
Brief Title: Reducing the Burden of Malaria by Targeting Hotspots of Malaria Transmission
Acronym: REDHOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other); Kenya Medical Research Institute (Other); Centers for Disease Control and Prevention (U.S. Federal Agency); International Centre of Insect Physiology and Ecology (ICIPE) (Other); Division of Malaria Control, Ministry of Health, Nairobi, Kenya (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: REDHOT_OPP1024438
Record Dates: First submitted 2012-03-19; First posted 2012-04-11 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Malaria
Keywords: malaria; heterogeneity; transmission; elimination
MeSH Terms: conditions — Malaria | interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hotspot Targeting (Experimental): Four hotspot-targeted interventions will be superimposed on ongoing control measures: hotspots will be targeted with a combination of IRS, long-lasting insecticide treated nets (LLINs), larviciding and a focal screening and treatment (FSAT)campaign.
  Interventions: Drug: Artemether-lumefantrine combination; Biological: Bacillus thuringiensis; Biological: Long lasting insecticide treated net (LLINs); Biological: Indoor Residual Spraying (IRS)
- Control (No Intervention): Standard of care as determined by the Division of Malaria Control of the Kenyan Ministry of Health

INTERVENTIONS:
Drug: Artemether-lumefantrine combination — Focal screening and treatment in all households in malaria hotspots prior to the peak transmission season. Screening of a sentinel age group by rapid diagnostic tests; all parasitaemic individuals and household members of parasitaemic individuals will be treated.
  Arms: Hotspot Targeting
Biological: Bacillus thuringiensis — Treatment of all waterbodies within hotspots with Bti or Bs on weekly basis
  Arms: Hotspot Targeting
Biological: Long lasting insecticide treated net (LLINs) — Distribution of LLINs in all households in malaria hotspots; instruction about correct use.
  Arms: Hotspot Targeting
Biological: Indoor Residual Spraying (IRS) — 6-monthly IRS with deltamethrin in all households malaria hotspots.
  Arms: Hotspot Targeting

SUMMARY:
In this study, the investigators propose to determine the value of rolling out four targeted malaria control efforts in reducing overall malaria transmission. These targeted control efforts include local upscaling of IRS and ITNs in hotspots of malaria transmission. In addition, larviciding will be employed to target malaria vectors, also those that are less susceptible to IRS and ITNs as a consequence of outdoor feeding and resting. Lastly, the human infectious reservoir will be reduced in hotspots of malaria transmission by treating parasite carriers and their household members with the current first-line antimalarial drug. The impact of these targeted interventions on overall transmission intensity will be assessed in the context of currently ongoing malaria control activities in a plausibility study. Hotspots of malaria transmission are defined in an area of 100km2 and randomized to receive hotspot targeted interventions and compared with their baseline and with control clusters where the routine (untargeted) malaria control activities continue. The interventions will be evaluated based on changes in parasite prevalence measured in community surveys inside and outside hotspots of malaria transmission. Parasite prevalence will be compared before and after the intervention in intervention clusters and between intervention and control clusters.

In addition to malaria surveys in the human population, an entomological evaluation will take place where the densities of mosquito larvae and adult mosquitoes are monitored longitudinally.

DETAILED DESCRIPTION:
DEFINITIONS This study uses a plausibility design to determine the plausible impact of hotspot-targeted interventions on overall malaria transmission. Hotspots will be detected in the 100km2 study area. Hotspots are defined as areas with a level of transmission intensity that exceeds that in the surrounding area; indicated by a higher sero-conversion rate and/or age-adjusted density of malaria-specific antibodies.

Clusters for the intervention are defined as a hotspot and the area surrounding this hotspot in each direction up to 500 meters.

INTERVENTION Half of the clusters will be randomized to hotspot-targeted interventions, while the other half will serve as control. The plausible impact of hotspot targeted interventions will be evaluated by comparing malaria indices in intervention clusters with their baseline and with control clusters.

In each phase four hotspot-targeted interventions will be superimposed on ongoing control measures: hotspots will be targeted with a combination IRS, long-lasting insecticide treated nets (LLINs), larviciding and a focal screening and treatment (FSAT).

EVALUATION The primary outcome will be parasite prevalence in evaluation zones (i.e. the area surrounding malaria hotspots) of targeted and untargeted clusters. In addition, parasite prevalence will be determined inside hotspots of malaria transmission and in evaluation zones in relation to distance to the hotspot boundary. For this, community surveys are planned prior to the intervention and at two time-points after the intervention.

An entomological evaluation will take place concurrently in which mosquito breeding sites are monitored for productivity and mosquitoes will be sampled indoors and outdoors.

Malaria morbidity is assessed by passive case detection.

ELIGIBILITY:
Exclusion Criteria:

* For LLINs, IRS and larviciding there are no exclusion criteria
* Pregnant women and children < 6 months of age are excluded from FSAT

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 17506 (Actual)
Dates: Start 2012-04; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Parasite prevalence in the evaluation zone surrounding malaria hotspots | 3 cross-sectional surveys in up to 210 days, the timing being: at enrolment; 45-75 days post enrolment (coinciding with the peak malaria transmission season) and 150-210 days post enrolment (coinciding with the end of the malaria transmission season)
  Parasite prevalence, determined by PCR, in the evaluation zone surrounding hotspots in intervention and control clusters

SECONDARY OUTCOMES:
Parasite prevalence inside malaria hotspots | 3 cross-sectional surveys in up to 210 days, the timing being: at enrolment; 45-75 days post enrolment (coinciding with the peak malaria transmission season) and 150-210 days post enrolment (coinciding with the end of the malaria transmission season)
  Parasite prevalence, determined by PCR, inside hotspot of malaria transmission in intervention and control clusters
Parasite prevalence in the evaluation zone as function of distance to the hotspot boundary | 3 cross-sectional surveys in up to 210 days, the timing being: at enrolment; 45-75 days post enrolment (coinciding with the peak malaria transmission season) and 150-210 days post enrolment (coinciding with the end of the malaria transmission season)
  Parasite prevalence, determined by PCR, in relation to distance to the boundary of malaria hotspots in intervention and control clusters
Anopheles mosquito density | determined during fortnightly trapping, starting at enrolment and continuing until up to 210 days after enrolment
  Indoor and outdoor anopheles mosquito density inside and outside hotspots of malaria transmission in intervention and control clusters
Passive case detection | determined continuously for a period of up to 210 days after enrolment
  Number of malaria cases reporting at health facilities, coming from intervention and control clusters
Safety and acceptability of interventions | at a single cross-sectional survey 15-45 days after enrolment
  Side effects of FSAT, LLINs and IRS in targeted households
Mosquito breeding site productivity | determined on a weekly basis for a period of up to 210 days after enrolment
  The presence and density of anopheles larvae in mosquito breeding sites in malaria hotspots in intervention and control clusters

CONTACTS AND LOCATIONS:
Overall Officials: Teun Bousema, PhD, Principal Investigator — Radboud University Medical Center; Jon Cox, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine; Jennifer Stevenson, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Rachuonyo District, Kenya

REFERENCES:
- [Background] Bousema T, Griffin JT, Sauerwein RW, Smith DL, Churcher TS, Takken W, Ghani A, Drakeley C, Gosling R. Hitting hotspots: spatial targeting of malaria for control and elimination. PLoS Med. 2012 Jan;9(1):e1001165. doi: 10.1371/journal.pmed.1001165. Epub 2012 Jan 31. PMID 22303287
- [Derived] Bousema T, Stresman G, Baidjoe AY, Bradley J, Knight P, Stone W, Osoti V, Makori E, Owaga C, Odongo W, China P, Shagari S, Doumbo OK, Sauerwein RW, Kariuki S, Drakeley C, Stevenson J, Cox J. The Impact of Hotspot-Targeted Interventions on Malaria Transmission in Rachuonyo South District in the Western Kenyan Highlands: A Cluster-Randomized Controlled Trial. PLoS Med. 2016 Apr 12;13(4):e1001993. doi: 10.1371/journal.pmed.1001993. eCollection 2016 Apr. PMID 27071072
- [Derived] Bousema T, Stevenson J, Baidjoe A, Stresman G, Griffin JT, Kleinschmidt I, Remarque EJ, Vulule J, Bayoh N, Laserson K, Desai M, Sauerwein R, Drakeley C, Cox J. The impact of hotspot-targeted interventions on malaria transmission: study protocol for a cluster-randomized controlled trial. Trials. 2013 Feb 2;14:36. doi: 10.1186/1745-6215-14-36. PMID 23374910